CLINICAL TRIAL: NCT07318090
Title: Developing a Family-Focused Treatment for Prolonged Grief for Parental Suicide Bereaved Families With Children
Brief Title: F-PGT - Prolonged Grief Treatment for Families Affected by Suicide
Acronym: F-PGT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American Foundation for Suicide Prevention (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Nadine Melhem, Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY23070021 (Aim 3); LSRG-0-080-22 (Other Grant/Funding Number: American Foundation for Suicide Prevention (AFSP))
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Prolonged Grief Disorder (PGD)
Keywords: Prolonged Grief Disorder; Suicide loss survivor; Family treatment; Prolonged Grief Treatment; Grief
MeSH Terms: conditions — Prolonged Grief Disorder

STUDY DESIGN:
Intervention Model Description: Open trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- F-PGT (Experimental): Eligible families will receive 16 online sessions of Family-Prolonged Grief Treatment (F-PGT).
  Interventions: Behavioral: F-PGT

INTERVENTIONS:
Behavioral: F-PGT — Family- Prolonged Grief Treatment (F-PGT) is a specialized talk therapy to help families who have lost a parent to suicide. It is based on Prolonged Grief Therapy (PGT) that is efficacious for adults and is now adapted for parents and their children ages 8 to 14. The therapy includes 16 online sessions where a therapist meets with the parent alone, the child alone, or both together. Activities for children are designed to match their age and understanding. The therapy guides families through six steps: understanding and accepting grief, seeing promise in the future, strengthening relationships, sharing the story of the death, living with reminders, and connecting with memories. As a part of the focus on strengthening relationships parents are encouraged to invite a friend or relative to join a session.

SUMMARY:
This pilot open trial is being done to better understand the needs of families who have lost a parent to suicide at least a year ago and who have children ages 8-14 and to develop and test Family-Prolonged Grief Treatment (F-PGT), a modification of prolonged grief therapy (PGT) as a way to help these families. PGT has been proven efficacious for adults with prolonged grief. The therapy has been adapted to include work with parents in helping their children (aged 8-14) and to include sessions with the child. All assessment and treatment sessions of the study are being conducted virtually.

DETAILED DESCRIPTION:
Interested potential adult participants will first complete a preliminary screening conducted by phone or secure zoom. Eligible and interested families will meet with a study clinician to provide written informed consent and child assent to participate in a 2-step study process. Step 1 is baseline assessment and confirming study eligibility, and step 2 is Prolonged Grief Treatment for Families (F-PGT).

Families who give consent will complete assessments to confirm eligibility for the study. Those who are not eligible will conclude their study participation. Eligible families will complete the remaining baseline assessments and proceed to step 2, treatment.

F-PGT includes 16 virtual sessions where a therapist will meet with either the parent or child, or both. All sessions will be recorded to continue optimize the therapy.

In addition, participants will complete regular assessments.

ELIGIBILITY:
Inclusion Criteria:

* Parental suicide bereaved children aged 8-14 years and their parents or caregivers.
* Child score of 68 or higher on the Inventory for Complicated Grief-Revised for Children (ICG-RC) and/or parent score of 5 or higher on the Brief Grief Questionnaire at phone screen and score of 30 or higher on the Inventory for Complicated Grief (ICG) at baseline.
* At least 12 months after death.
* Child and/or parent's primary concern is prolonged grief
* Child has a biological/adoptive parent or court-appointed guardian who can present paperwork that they are able to consent for research for the youth involved in the study. Child is currently living with this caregiver and has spent most of their time in the past year under their care.
* Both child and parent/caregiver have a clinical provider to communicate safety concerns (e.g., primary care provider, pediatrician)
* Both child and parent/caregiver live in the United States
* If taking psychoactive medications, has been on a stable dose for at least 3 months.

Exclusion Criteria:

Youth exclusion criteria:

* Limited cognitive abilities to assent or to participate in the therapy (e.g., acute mania, psychosis, severe autism spectrum disorder)
* Unstable serious medical condition
* Current residence is in a state in which none of the study therapists are licensed (i.e., Alaska, Hawaii, Iowa, Louisiana, Massachusetts, Montana, New Mexico, Oregon)
* Has a substance use disorder (determined by KSADS during the baseline assessment)
* Is currently in therapy or begins therapy during the period of study participation
* Those with active suicidality (C-SSRS scores of 3 or higher)
* Those who report any suicidal behaviors in the past year (i.e., suicide attempt, interrupted attempt, aborted attempt, preparatory behaviors), including any formal crisis management in the past year (e.g., presented at emergency department for suicidality), as assessed at baseline.

Parent/Caregiver Exclusion criteria:

* Age younger than 18 years old
* Limited cognitive abilities to consent (e.g., acute mania, psychosis)
* Unstable serious medical condition
* For those with active suicidality (C-SSRS scores of 3 or higher), eligibility will be determined by the clinical team and PIs based on prior history of suicidality, access to lethal means, availability social support, reasons for living, and engagement in safety planning.
* Those who report any suicidal behaviors in the past year (i.e., suicide attempt, interrupted attempt, aborted attempt, preparatory behaviors), including any formal crisis management in the past year (e.g., presented at emergency department for suicidality), as assessed at baseline.
* Is currently in therapy or begins therapy during the study duration
* Current residence is in a state in which none of the study therapists are licensed (i.e., Alaska, Hawaii, Iowa, Louisiana, Massachusetts, Montana, New Mexico, Oregon)
* Has a substance use disorder (determined by SCID during the baseline assessment)

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total Score on Feasibility of Intervention Measure (FIM) at End of Treatment | End of treatment at 20 weeks
  Total scores from the Feasibility of Intervention Measure (FIM) will be used to assess participants' perception of intervention feasibility. Total Score FIM: 4-8 Low feasibility; 9-15 Moderate feasibility; 16-20 High feasibility.
Total Score on Acceptability of Intervention Measure (AIM) at End of Treatment | End of treatment at 20 weeks
  Total scores from the Acceptability of Intervention Measure (AIM) will be used to assess participants' perception of intervention acceptability. Total Score AIM: 4-8 Low acceptability; 9-15 Moderate acceptability; 16-20 High acceptability.
Change in Inventory of Complicated Grief (ICG) Total Score | Baseline; 4, 8, 12, and 16 weeks of treatment; 20 weeks assessment
  Total scores from the Inventory of Complicated Grief (ICG) will be used to assess severity of complicated grief symptoms in adults. Total Score ICG: 0-24 Minimal grief; 25-29 Mild/moderate grief; ≥30 Clinically significant grief.
Change in Inventory for Complicated Grief-Revised for Children (ICG-RC) Total Score | Baseline; 4, 8, 12, and 16 weeks of treatment; 20 weeks assessment
  Total scores from the Inventory for Complicated Grief-Revised for Children (ICG-RC) will be used to assess severity of prolonged grief symptoms in children and adolescents. Total Score ICG-RC: 28-67 Minimal/mild grief; ≥68 Clinically significant prolonged grief.
Change in Clinical Global Impression (CGI-S and CGI-I) Scores | Baseline; 4, 8, 12, and 16 weeks of treatment; 20 weeks assessment
  Clinician-rated scores from the Clinical Global Impression scale will be used to assess global severity and improvement. CGI-Severity: 1-2 Normal/mild; 3-4 Moderate; 5-7 Severe. CGI-Improvement: 1-2 Improved; 3-4 No change; 5-7 Worsened.

SECONDARY OUTCOMES:
Change in Child Global Assessment Scale (C-GAS) Total Score | Baseline; 4, 8, 12, and 16 weeks of treatment; 20 weeks assessment
  Total scores from the Children's Global Assessment Scale (C-GAS) will be used to assess overall child functioning. Total Score C-GAS: 91-100 Superior functioning; 71-90 Good functioning; 51-70 Moderate impairment; 31-50 Serious impairment; 1-30 Severe impairment.
Change in Global Assessment Scale (GAS) Total Score (Parent) | Baseline; 4, 8, 12, and 16 weeks of treatment; 20 weeks assessment
  Total scores from the Global Assessment Scale (GAS) will be used to assess overall parental functioning. Higher scores indicate better functioning.
Change in Work and Social Adjustment Scale (WSAS) Total Score | Baseline; 4, 8, 12, and 16 weeks of treatment; 20 weeks assessment
  Total scores from the Work and Social Adjustment Scale (WSAS) will be used to assess functional impairment. Total Score WSAS: 0-9 Low impairment; 10-20 Significant impairment; >20 Moderately severe to severe impairment.
Change in Parental Reflective Functioning Questionnaire (PRFQ) Total Score | Baseline; 4, 8, 12, and 16 weeks of treatment; 20 weeks assessment
  Total scores from the Parental Reflective Functioning Questionnaire (PRFQ) will be used to assess parents' capacity to reflect on their child's mental states. Higher scores indicate greater reflective functioning, except for the Pre-mentalizing subscale where higher scores indicate less adaptive functioning.
Change in Coping with Children's Negative Emotions Scale (CCNES) Total Score | Baseline; 20 weeks assessment
  Total scores from the Coping with Children's Negative Emotions Scale (CCNES) will be used to assess parental responses to children's negative emotions. Higher supportive response scores reflect more adaptive parenting.
Change in Child and Adolescent Reflective Functioning Scale (CARFS) Score | Baseline; 4, 8, 12, and 16 weeks of treatment; 20 weeks assessment
  Total scores from the Child and Adolescent Reflective Functioning Scale (CARFS) will be used to assess children's ability to understand their own and others' mental states. Higher scores indicate greater reflective functioning.
Change in Child-Parent Relationship Scale (CPRS) Total Score | Baseline; 4 weeks; 12 weeks; 20 weeks assessment
  Total scores from the Child-Parent Relationship Scale (CPRS) will be used to assess parent-child relationship quality. Higher scores indicate more positive relationship quality or greater stress on stress-related subscales.
Presence of Psychiatric Diagnoses as Assessed by Structured Clinical Interview for DSM-5 (SCID-5) | Baseline
  Diagnostic outcomes from the Structured Clinical Interview for DSM-5 (SCID-5) will be used to assess the presence of DSM-5 psychiatric disorders in adults for inclusion/exclusion criteria and will help in assessing global functioning. Each disorder will be coded as 0 (not present), 1 (subthreshold), or 2 (present).
Change in Psychiatric Diagnoses as Assessed by Structured Clinical Interview for DSM-5 (SCID-5) | End of treatment at 20 weeks
  Diagnostic outcomes from the Structured Clinical Interview for DSM-5 (SCID-5) will be used to assess changes in DSM-5 psychiatric disorders in adults and in global functioning. Each disorder will be coded as 0 (not present), 1 (subthreshold), or 2 (present).
Presence of Psychiatric Diagnoses as Assessed by K-SADS-PL (Child and Parent Versions) | Baseline; 20 weeks assessment
  Diagnostic outcomes from the Kiddie Schedule for Affective Disorders and Schizophrenia - Present and Lifetime Version (K-SADS-PL) will be used to assess DSM psychiatric disorders in children and adolescents for inclusion/exclusion criteria and will help in assessing global functioning. Each disorder will be coded as 1 (not present), 2 (subthreshold), or 3 (present).
Change in DSM Psychiatric Diagnoses as Assessed by Kiddie Schedule for Affective Disorders and Schizophrenia - Present and Lifetime Version (K-SADS-PL) | End of treatment at 20 weeks
  Diagnostic outcomes from the Kiddie Schedule for Affective Disorders and Schizophrenia - Present and Lifetime Version (K-SADS-PL) will be used to assess changes in DSM psychiatric disorders in children and adolescents and in global functioning. Each disorder will be coded as 1 (not present), 2 (subthreshold), or 3 (present).
Total Score on Prolonged Grief Disorder-13 (PG-13) Scale | Baseline
  Total scores from the Prolonged Grief Disorder-13 (PG-13) scale will be used to assess severity of prolonged grief symptoms. Total Score PG-13: 10-29 Mild grief; 30-50 Clinically significant prolonged grief.
Change in Total Score on Prolonged Grief Disorder-13 (PG-13) Scale | 20 weeks assessment
  Total scores from the Prolonged Grief Disorder-13 (PG-13) scale will be used to assess severity of prolonged grief symptoms. Total Score PG-13: 10-29 Mild grief; 30-50 Clinically significant prolonged grief.
Observed Parent-Child Communication Behaviors During Virtual Interaction Tasks | Baseline
  Observed parent-child communication behaviors will be assessed during three 5-minute structured virtual interaction tasks (discussion of friendships, resolution of a minor conflict, and planning a "dream vacation"). Video-recorded sessions will be coded by trained raters using a standardized observational coding system. Higher scores indicate more adaptive communication behaviors.
Change in Observed Parent-Child Communication Behaviors During Virtual Interaction Tasks | End of treatment at 20 weeks
  Change in observed parent-child communication behaviors will be assessed during three 5-minute structured virtual interaction tasks. Video-recorded sessions will be coded by trained raters using a standardized observational coding system. Positive change scores indicate improvement in communication behaviors from baseline.
Observed Parent-Child Attachment Behaviors During Virtual Interaction Tasks | Baseline
  Observed attachment-related behaviors between parent and child will be assessed during three 5-minute structured virtual interaction tasks. Video-recorded sessions will be coded by trained raters using a standardized observational coding system. Higher scores indicate more secure attachment behaviors.
Change in Observed Parent-Child Attachment Behaviors During Virtual Interaction Tasks | End of treatment at 20 weeks
  Change in observed parent-child attachment behaviors will be assessed during three 5-minute structured virtual interaction tasks. Video-recorded sessions will be coded by trained raters using a standardized observational coding system. Positive change scores indicate improvement in attachment behaviors from baseline.
Observed Parent and Child Reflective Functioning During Virtual Interaction Tasks | Baseline
  Observed reflective functioning of parents and children will be assessed during three 5-minute structured virtual interaction tasks. Video-recorded sessions will be coded by trained staff using a validated reflective functioning coding framework. Higher scores indicate greater capacity to recognize and interpret mental states.
Change in Observed Parent and Child Reflective Functioning During Virtual Interaction Tasks | End of treatment at 20 weeks
  Change in observed reflective functioning of parents and children will be assessed during three 5-minute structured virtual interaction tasks. Video-recorded sessions will be coded by trained staff using a validated reflective functioning coding framework. Positive change scores indicate improvement in reflective functioning from baseline.

OTHER OUTCOMES:
Change in Depressive Symptoms as Assessed by Quick Inventory of Depressive Symptomatology (QIDS) | Baseline; 12 weeks; 20 weeks assessment
  Total scores from the Quick Inventory of Depressive Symptomatology (QIDS) will be used to assess depressive symptom severity. Higher scores indicate greater depression severity.
Change in Anxiety Symptoms as Assessed by Generalized Anxiety Disorder-7 (GAD-7) | Baseline; 12 weeks; 20 weeks assessment
  Total scores from the Generalized Anxiety Disorder-7 (GAD-7) will be used to assess anxiety severity. Higher scores indicate greater anxiety.
Change in Posttraumatic Stress Symptoms as Assessed by Davidson Trauma Scale (DTS) | Baseline; 12 weeks; 20 weeks assessment
  Total scores from the Davidson Trauma Scale (DTS) will be used to assess severity of posttraumatic stress symptoms. Higher scores indicate greater trauma-related distress.
Change in Child Anxiety and Depression Symptoms as Assessed by RCADS-25 (Child and Parent Versions) | Baseline; 12 weeks; 20 weeks assessment
  Total scores from the Revised Children's Anxiety and Depression Scale - Short Version (RCADS-25) will be used to assess anxiety and depressive symptoms in children and adolescents. Higher scores indicate greater symptom severity.
Suicidal Ideation and Behavior as Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline; weekly during treatment; 20 weeks assessment
  Scores from the Columbia-Suicide Severity Rating Scale (C-SSRS) will be used to assess severity and frequency of suicidal ideation and behavior in adults and children. The C-SSRS ideation severity subscale is scored on a 5-point ordinal scale ranging from 1 (wish to be dead) to 5 (active suicidal ideation with specific plan and intent), with higher scores indicating greater severity of suicidal ideation and a worse clinical outcome.
Change in Family Functioning as Assessed by Family Adaptability and Cohesion Scale (FACES-IV-SF) | Baseline; 12 weeks; 20 weeks assessment
  Total scores from the Family Adaptability and Cohesion Scale - Short Form (FACES-IV-SF) will be used to assess family functioning. Higher scores indicate healthier family dynamics.
Change in Parenting Competence as Assessed by Parenting Sense of Competency Scale (PSCS) | Baseline; 12 weeks; 20 weeks assessment
  Total scores from the Parenting Sense of Competency Scale (PSCS) will be used to assess parental efficacy and satisfaction. Higher scores indicate greater perceived parenting competence.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine A Melhem, PhD, Principal Investigator — University of Pittsburgh; M. Katherine Shear, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Not required by the funding agency.

REFERENCES:
- [Background] Melhem NM, Walker M, Moritz G, Brent DA. Antecedents and sequelae of sudden parental death in offspring and surviving caregivers. Arch Pediatr Adolesc Med. 2008 May;162(5):403-10. doi: 10.1001/archpedi.162.5.403. PMID 18458185
- [Background] Melhem NM, Porta G, Shamseddeen W, Walker Payne M, Brent DA. Grief in children and adolescents bereaved by sudden parental death. Arch Gen Psychiatry. 2011 Sep;68(9):911-9. doi: 10.1001/archgenpsychiatry.2011.101. PMID 21893658
- [Background] Hamdan S, Mazariegos D, Melhem NM, Porta G, Payne MW, Brent DA. Effect of parental bereavement on health risk behaviors in youth: a 3-year follow-up. Arch Pediatr Adolesc Med. 2012 Mar;166(3):216-23. doi: 10.1001/archpediatrics.2011.682. PMID 22393180
- [Background] Pham S, Porta G, Biernesser C, Walker Payne M, Iyengar S, Melhem N, Brent DA. The Burden of Bereavement: Early-Onset Depression and Impairment in Youths Bereaved by Sudden Parental Death in a 7-Year Prospective Study. Am J Psychiatry. 2018 Sep 1;175(9):887-896. doi: 10.1176/appi.ajp.2018.17070792. Epub 2018 Jun 20. PMID 29921145
- [Background] Melhem NM, Porta G, Walker Payne M, Brent DA. Identifying prolonged grief reactions in children: dimensional and diagnostic approaches. J Am Acad Child Adolesc Psychiatry. 2013 Jun;52(6):599-607.e7. doi: 10.1016/j.jaac.2013.02.015. Epub 2013 Apr 24. PMID 23702449
- [Background] Melhem NM, Moritz G, Walker M, Shear MK, Brent D. Phenomenology and correlates of complicated grief in children and adolescents. J Am Acad Child Adolesc Psychiatry. 2007 Apr;46(4):493-499. doi: 10.1097/chi.0b013e31803062a9. PMID 17420684
- [Background] Shear K, Frank E, Houck PR, Reynolds CF 3rd. Treatment of complicated grief: a randomized controlled trial. JAMA. 2005 Jun 1;293(21):2601-8. doi: 10.1001/jama.293.21.2601. PMID 15928281
- [Background] Shear MK, Wang Y, Skritskaya N, Duan N, Mauro C, Ghesquiere A. Treatment of complicated grief in elderly persons: a randomized clinical trial. JAMA Psychiatry. 2014 Nov;71(11):1287-95. doi: 10.1001/jamapsychiatry.2014.1242. PMID 25250737
- [Background] Shear MK, Reynolds CF 3rd, Simon NM, Zisook S, Wang Y, Mauro C, Duan N, Lebowitz B, Skritskaya N. Optimizing Treatment of Complicated Grief: A Randomized Clinical Trial. JAMA Psychiatry. 2016 Jul 1;73(7):685-94. doi: 10.1001/jamapsychiatry.2016.0892. PMID 27276373
- [Background] Hamdan S, Melhem NM, Porta G, Song MS, Brent DA. Alcohol and substance abuse in parentally bereaved youth. J Clin Psychiatry. 2013 Aug;74(8):828-33. doi: 10.4088/JCP.13m08391. PMID 24021502